CLINICAL TRIAL: NCT03891602
Title: Using a Mixed Methods Approach to Understand Shared Decision-Making in Lung Cancer Screening
Brief Title: DECIDE: Developing Tools for Lung Cancer Screening Discussion Improvement
Acronym: DECIDE
Status: Completed | Type: Observational
Sponsor: Hackensack Meridian Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Indiana University (Other); University of North Carolina (Other); Memorial Sloan Kettering Cancer Center (Other); Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Lisa Carter-Bawa, PhD, Director | Cancer Prevention Precision Control Institute, Hackensack Meridian Health
Other Study IDs: 19-007; Pro2022-0776 (Other: Hackensack Meridian Health IRB)
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Smoking; Smoking, Tobacco; Smoking, Cigarette; Lung Cancer
Keywords: Smoker; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Smoking; Tobacco Smoking; Cigarette Smoking; Lung Neoplasms | interventions — Cycloserine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinicians: Primary care clinicians (general internists, family physicians, nurse practitioners, physician assistants) who treat lung cancer screening eligible patients
  Interventions: Behavioral: Primary Care Clinicians' Lung Cancer Screening Survey
- Smokers/Former Smokers: Current smoker or former smoker who has quit within the past 15 years
  Interventions: Behavioral: Cataldo Lung Cancer Stigma Scale (Smoking-Related Subscale); Behavioral: Patient Trust in the Medical; Behavioral: Decision Conflict Scale (DCS) - Lung Cancer Screening; Behavioral: Shared Decision Making Questionnaire (SDM-Q)- Patient; Behavioral: Stage of Readiness for Smoking Cessation - Contemplation Ladder

INTERVENTIONS:
Behavioral: Cataldo Lung Cancer Stigma Scale (Smoking-Related Subscale) — Perceived Smoking-Related Stigma will be measured using the 5-item Cataldo Lung Cancer Stigma Scale (Smoking-Related Subscale). The response scale is 1 = strongly disagree, to 4 = strongly agree, and scores range from 5 to 25 (high stigma). Cronbach's alphas were 0.75 to 0.89 in prior studies.
  Groups: Smokers/Former Smokers
Behavioral: Patient Trust in the Medical — Medical Mistrust will be measured using the 5-item Patient Trust in the Medical Profession Scale.80 The five-point Likert responses measure the extent to which patients perceive their clinician to be honest, caring more about convenience, thorough and careful, and trusted. The range of scores is 5 to 25 (higher mistrust). Reliability and validity have been well established with a Cronbach"s alpha of 0.84.
  Groups: Smokers/Former Smokers
Behavioral: Decision Conflict Scale (DCS) - Lung Cancer Screening — The DCS is a 16-item Likert-response item scale that has been modified for the lung cancer screening and smoking cessation contexts. The DCS was developed by O"Connor,74-75 and validated in many health decisions including breast cancer screening with Cronbach"s alphas ranging from 0.78 to 0.81. 74-75 Despite its name, the DCS measures more than decision conflict to encompass personal perceptions of perceived decision-making quality such as feeling the choice is informed, values based, and likely to be implemented as well as expressing satisfaction with the decision. 74-75 The DCS is comprised of items with response options ranging from 1 (strongly disagree) to 5 (strongly agree). The items are summed to total scale score with lower scores reflective of higher decision conflict and higher scores reflective of lower decision conflict.
  Other Names: DCS
  Groups: Smokers/Former Smokers
Behavioral: Shared Decision Making Questionnaire (SDM-Q)- Patient — Shared Decision Making Process will be measured from the patient perspective using the 9-item Shared Decision Making Questionnaire (SDM-Q-9),77 which has been validated with a Cronbach"s alpha of 0.94.
  Other Names: SDM-Q-9
  Groups: Smokers/Former Smokers
Behavioral: Stage of Readiness for Smoking Cessation - Contemplation Ladder — Among current smokers
  Groups: Smokers/Former Smokers
Behavioral: Primary Care Clinicians' Lung Cancer Screening Survey — Includes items to assess attitudes, barriers, and knowledge of lung cancer screening guidelines.
  Groups: Clinicians

SUMMARY:
The purpose of this study is to learn about discussion between clinicians and their patients related to lung screening. Survey answers will be collected from both clinicians and their patients.

ELIGIBILITY:
Inclusion Criteria:

CLINICIANS:

* Clinician (physician, nurse practitioner, or physician assistant)
* Practicing in a KPWA primary care clinic
* Having a patient panel with >/= 10 lung cancer screening eligible patients

PATIENTS (Quantitative Phase):

* Age 55-80 years
* >/= 30 pack-year tobacco smoking history
* Current smoker or former smoker who has quit within the past 15 years
* Documented SDM lung cancer screening discussion during a recent clinic visit

Exclusion Criteria:

PATIENTS:

* Significant comorbidities (Charlson Comorbidity Index >/=3)
* Lung cancer diagnosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All recruitment will take place at Kaiser Permanente Washington.
Sampling Method: Probability Sample
Enrollment: 654 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Ostroff, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Lisa Carter-Bawa, PhD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Kaiser Permanente Washington Health Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
• Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clinicians | Smokers/Former Smokers
Started | 125 | 529
Completed | 125 | 529
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Clinicians and patients included in the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinicians | Smokers/Former Smokers | Total
Number analyzed (Participants) | 125 | 529 | 654
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Clinicians who participated in the study were only asked for their age as a categorical variable as a result we cannot provide mean and standard deviation.
  years
    number analyzed (Participants) | 0 | 529 | 529
    (all) |  | 66.4 (5.9) | 66.4 (5.9)
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0
  ≥ 18 and ≤ 50 years | 80 | 0 | 80
  > 50 years | 45 | 529 | 574
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 81 | 235 | 316
  Male | 43 | 294 | 337
  Prefer not to say | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 12 | 17
  Not Hispanic or Latino | 120 | 517 | 637
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 21 | 23 | 44
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 14 | 16
  White | 79 | 463 | 542
  More than one race | 7 | 9 | 16
  Unknown or Not Reported | 13 | 17 | 30
Region of Enrollment [Number; unit: participants]
  United States | 125 | 529 | 654

OUTCOME MEASURES:

1. Primary Outcome: Key Components of Shared Decision Making Process That Predict Patient-perceived Lung Cancer Screening Decision Quality
Description: Decisional Quality was measured using the multidimensional Decisional Conflict Scale, a 16-item Likert-response scale that was modified by the investigators for the lung cancer screening context. The total score ranging from 0 to 64. This total score is commonly transformed into a standardized score that falls within a 0 to 100 range. Decisional quality measured on this numeric scale from which lower scores represent lower decisional conflict and, therefore, higher decisional quality. Scores below 25 have been associated with low decisional conflict.
Time Frame: at baseline (study enrollment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smokers/Former Smokers
Number analyzed (Participants) | 529
score on a scale | 21.5 (15.5)

ADVERSE EVENTS:
Time Frame: Within 12 months
Description: Self reported adverse events
Arm/Group | Clinicians | Smokers/Former Smokers
All-Cause Mortality (participants affected / at risk) | 0/125 | 0/529
Serious Adverse Events (participants affected / at risk) | 0/125 | 0/529
Other Adverse Events (participants affected / at risk) | 0/125 | 0/529

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/02/NCT03891602/Prot_SAP_000.pdf